CLINICAL TRIAL: NCT02343081
Title: A Randomized, Open Label, Two-way Crossover, Single Dose Bioequivalence Study Comparing Dralitem® Capsules to the Reference Drug Temodal® Capsules in Patients With Primary Tumors of the Central Nervous System Under Fasting Conditions
Brief Title: Bioequivalence Study of Temozolomide in Patients With Primary Tumors of the Central Nervous System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Monte Verde SA (Industry)
Collaborators: FLENI Instituto de Rehabilitación y Educación Terapéutica, BA, Argentina. (Unknown); Bioanalytical Unit, Laboratorio Raffo S.A., BA, Argentina. (Unknown); FLENI Multi-Specialty Research Center, BA, Argentina. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RFF -0208
Record Dates: First submitted 2015-01-07; First posted 2015-01-21 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Brain Neoplasms, Malignant, Primary
Keywords: brain neoplasm; bioequivalence; temozolomide
MeSH Terms: conditions — Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temodal (Active Comparator): Temozolomide (Schering-Plough) 200 mg/m2, single oral dose.
  Interventions: Drug: Temozolomide
- Dralitem (Experimental): Temozolomide (Monte Verde S.A.) 200 mg/m2, single oral dose
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodal
  Arms: Temodal
Drug: Temozolomide
  Other Names: Dralitem
  Arms: Dralitem

SUMMARY:
The purpose of this crossover, single-dose, bioequivalence study is to compare the rate and extent of absorption of Temozolomide after the administration of the study product (Dralitem®, Monte Verde S.A.) and the reference product (Temodal®, Schering Plough) in primary Central Nervous System patients.

DETAILED DESCRIPTION:
Prospective, randomized, two-period, two treatment, two-way crossover bioequivalence study of two Temozolomide oral formulations (Dralitem vs. Temodal), in primary Central Nervous System tumor patients under fasting conditions. Open label to the patients and investigators and blind to the bioanalytical and clinical laboratories.

Study plan: days -21 to 0 (Recruitment period); days 1 to 5 (Treatment period); days 6 to 21 (Safety surveillance period). Sample size: 24 patients will be randomized. The patients will be administered Temozolomide 200 mg/m2 on the first two days (Dralitem) of the treatment cycle.

They will be admitted to the study clinical site on the evening of day 2. In the morning of day 3 they will be randomized into two groups of equal size. According to the assigned random number, each subject will receive a single oral dose of Temozolomide 200mg/m2 from either Monte Verde Sociedad Anónima (SA) product (Dralitem) or from Schering-Plough product (Temodal). The single dose of 200 mg/m2 will be reached with three different Temozolomide capsule strengths: 20, 100 and 250 mg. Drugs will be administered with 200-240 ml of water in semi-sitting upright position.

The following day (day 4) each subject will receive an oral dose of Temozolomide 200 mg/m2 of the product that did not receive the day before. On days 3 and 4 after drug administration, blood samples will be obtained for pharmacokinetic evaluation. The patient will be discharged from the clinical site on day 4 after completion of sampling for pharmacokinetic analysis. On day 5, all patients will receive Temozolomide 200 mg/m2 (Dralitem).

On days 3 and 4, samples of venous blood will be withdrawn from the forearm vein of each volunteer at the following time points: 0 (pre-dose) and 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours post-dose after each period administration. The washout period between the treatment arms was 10 hours, on days 3 and 4. Samples will be processed according to the validated method MANA (Método Analítico) - PLB (Proyecto Laboratorio Bioanalítico) 004 - TEM (Temozolomide) - 01/01. Measurement of plasma concentration of Temozolomide was performed using High Performance Liquid Chromatography (HPLC) followed by detection by tandem mass spectrometry (MS / MS).

The area under the curve (AUC) and the Cmax levels of the drug vs. time will be obtained for each subject. The resulting values of the logarithmic transformation of these parameters will be used for statistical comparisons (mixed effects ANOVA). The limits of the 90% confidence interval for the ratio of log transformed pharmacokinetic parameters will be calculated. Bioequivalence criteria: each calculated confidence interval should be within the acceptance range from 80.00 to 125.00.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with primary malignant tumors of the central nervous system (CNS) excluding subjects with primary CNS lymphoma.
2. Age> 21 years.
3. There should be a gap of two weeks between the last surgery and/or radiotherapy procedure and the day of randomization. If the procedure were intrabdominal, the gap should be of four weeks.
4. Patients with neutrophils> 1.5 x 109 / L and platelets> 100 x 109 / L.
5. Signed written informed consent for participation in the trial.

Exclusion Criteria:

1. Known hypersensitivity to Temozolomide or any other ingredient of the pharmaceutical formulation.
2. Any situation (eg. vomiting) that may interfere with the absorption of the product under study.
3. Chemotherapy or biological therapy within four weeks prior to administering the products under study.
4. Patients who experience any symptoms of toxicity to prior antineoplastic therapies upon administration of the products under study.
5. Participation in other clinical research studies during the 90 days before the start of this study.
6. History of alcohol or drugs abuse.
7. History of severe allergic reactions to any type of antigen.
8. History of gastrointestinal surgery (except uncomplicated appendectomy, of at least three months old).
9. Patients whose clinical status would affect the safety of the products under study or interfere with the pharmacokinetic evaluation, at the discretion of the investigator.
10. Pregnant women or women planning to become pregnant during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro D Muggeri, Physician, Principal Investigator — FLENI Instituto Clínico-Quirúrgico de Diagnóstico y Tratamiento
Locations (2):
- Argentina (2):
  - FLENI Instituto de Rehabilitación y Educación Terapéutica, Belén de Escobar, Buenos Aires
  - FLENI Instituto Clínico-Quirúrgico de Diagnóstico y Tratamiento, Ciudad Autónoma de Buenos Aires, Buenos Aires

REFERENCES:
- [Derived] Muggeri A, Vago M, Perez S, Rubio M, Gonzalez C, Magarinos C, Rosenberg M, Costa F, Perez-Lloret S. A Randomized, Open-Label, Two-Way Crossover, Single-Dose Bioequivalence Study of Temozolomide 200 mg/m2 (Dralitem(R) vs. Temodal(R) Capsules) in Patients with Primary Tumors of the Central Nervous System Under Fasting Conditions. Drugs R D. 2017 Sep;17(3):427-434. doi: 10.1007/s40268-017-0199-3. PMID 28756607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with primary tumours of the Central Nervous System (CNS) excluding patients with primary CNS lymphoma, from FLENI Clinical-Surgical Diagnosis and Treatment Institute, Buenos Aires, Argentina. The last patient completed in October 2013.
Pre-assignment Details: Of the initial sample size of 24 patients, 19 were effectively screened during a period from October 2012 and October 2013; 3 patients did not meet inclusion criteria and 16 were randomized to the two intervention arms.
Groups:
- Temodal, Then Dralitem: During days 1 and 2, all patients received a single oral dose of 200 mg/m2 of Temozolomide from Monte Verde S.A. (Dralitem®). On day 3 patients received 200 mg/m2 of Temozolomide from Schering-Plough (Temodal®) as a single oral dose. After a washout period of 10 hours, they then received 200 mg/m2 of Temozolomide from Monte Verde S.A. (Dralitem®). On day 5 all patients received Temozolomide 200 mg/m2 from Monte Verde S.A. (Dralitem®).All patients were under fasting conditions two hours before and after each drug administration.
- Dralitem, Then Temodal: During days 1 and 2, all patients received a single oral dose of 200 mg/m2 of Temozolomide from Monte Verde S.A. (Dralitem®). On day 3 patients received 200 mg/m2 of Temozolomide from Monte Verde S.A. (Dralitem®) as a single oral dose. After a washout period of 10 hours, they then received 200 mg/m2 of Temozolomide from Schering-Plough (Temodal®). On day 5 all patients received Temozolomide 200 mg/m2 from Monte Verde S.A.(Dralitem®). All patients were under fasting conditions two hours before and after each drug administration.
Period: First Intervention (Day 3)
Arm/Group | Temodal, Then Dralitem | Dralitem, Then Temodal
Started | 8 | 8
Received Intervention | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (10 Hours)
Arm/Group | Temodal, Then Dralitem | Dralitem, Then Temodal
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (Day 4)
Arm/Group | Temodal, Then Dralitem | Dralitem, Then Temodal
Started | 8 | 8
Received Intervention | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Temodal, Then Dralitem | Dralitem, Then Temodal | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.75 (9.35) | 39.75 (14.5) | 48.44 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Argentina | 8 | 8 | 16
Height [Mean (Standard Deviation); unit: cm] | 169 (9.53) | 173.37 (8.65) | 170.00 (8.00)
Weight, Continuous [Mean (Standard Deviation); unit: kg] | 78.87 (14.20) | 81.12 (10.78) | 79.40 (12.00)
Body Surface, Continuous [Mean (Standard Deviation); unit: m^2] | 1.89 (0.22) | 1.95 (0.16) | 1.92 (0.19)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.03 (2.01) | 28.46 (2.72) | 27.26 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Rate of absorption of Temozolomide (Cmax) will be measured after the oral administration of the test product (Dralitem®, Monte Verde S.A.) or the reference product (Temodal®, Schering-Plough).
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours on Days 3 and 4
Population: All those subjects who completed the study and were compliant with all the protocol procedures were considered evaluable for statistical pharmacokinetic analysis. Those who received at least one dose of the products under study but did not comply with the study procedures were included in the safety analysis only.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Temodal: Temozolomide (Schering-Plough) 200 mg/m2, single oral dose.
  Temozolomide
- Dralitem: Temozolomide (Monte Verde S.A.) 200 mg/m2, single oral dose
  Temozolomide
Arm/Group | Temodal | Dralitem
Number analyzed (Participants) | 16 | 16
mcg/mL | 11.108 (2.486) | 10.575 (2.805)
Statistical Analysis 1: Comparison: Temodal vs Dralitem; Bioequivalence assessment was made for the 90% CI for the ratio of log transformed pharmacokinetic parameters μT / μR and with the two one-sided Schuirmann T-test procedure under the null hypothesis; Test type: Non-Inferiority or Equivalence — Assuming an intrasubject CV of 15%, an enrollment of 16 subjects was selected to provide a minimum of 80% power for the 90% CI of the ratio of the mean for Cmax for Temozolomide reference and test to fall within the 80-125% confidence range; p < 0.05, ANOVA; Primary parameters were analyzed using ANOVA. A linear, mixed model for crossover designs (two-period, two-sequence, two-treatment) was used; Cmax = 94.37, 90% CI 2-sided [82.69 to 107.69] — Cmax Test/Reference Ratio

2. Secondary Outcome: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs and SAEs will be collected from the start of study treatment and until two weeks post last dose. If AEs or SAEs extend in time and are not resolved before the end of the 2-week follow up period, this period shall last until the event/s are resolved.
Time Frame: Up to two weeks post last dose
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Kel
Description: Rate at which Temozolomide is removed from the body.
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours on Days 3 and 4
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Temodal | Dralitem
Number analyzed (Participants) | 16 | 16
1/h | 0.3743 (0.0451) | 0.3691 (0.0258)

4. Other Pre Specified Outcome: T1/2
Description: Time required for Temozolomide plasma concentration to decrease by 50%
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours on Days 3 and 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Temodal | Dralitem
Number analyzed (Participants) | 16 | 16
hours | 1.87 (0.20) | 1.89 (0.13)

5. Primary Outcome: AUC0-t
Description: Extent of absorption of Temozolomide from time (0) to the last quantifiable concentration (t) will be measured after the oral administration of the test product (Dralitem®, Monte Verde S.A.) or the reference product (Temodal®, Schering-Plough)
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours on Days 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Temodal | Dralitem
Number analyzed (Participants) | 16 | 16
mcg*h/mL | 30.796 (3.893) | 31.104 (4.019)
Statistical Analysis 1: Comparison: Temodal vs Dralitem; Test type: Non-Inferiority or Equivalence — Assuming an intrasubject CV of 15%, an enrollment of 16 subjects was selected to provide a minimum of 80% power for the 90% CI of the means ratio for AUC0-t for Temozolomide reference and test to fall within the 80-125% confidence range; p < 0.05, ANOVA; AUC0-t = 100.99, 90% CI 2-sided [97.81 to 104.28] — AUC0-t Test/Reference Ratio

6. Primary Outcome: AUC0-∞
Description: Extent of absorption of Temozolomide from time (0) to infinity (∞) will be measured after oral administration of the test product (Dralitem®, Monte Verde S.A.) or the reference product (Temodal®, Schering-Plough).
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0 hours on Days 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Temodal | Dralitem
Number analyzed (Participants) | 16 | 16
mcg*h/mL | 31.817 (4.159) | 32.290 (4.174)
Statistical Analysis 1: Comparison: Temodal vs Dralitem; Test type: Non-Inferiority or Equivalence — Assuming an intrasubject CV of 15%, an enrollment of 16 subjects was selected to provide a minimum of 80% power for the 90% CI of the means ratio for AUC0-inf for Temozolomide reference and test to fall within the 80-125% confidence range; p < 0.05, ANOVA; AUC0-inf = 101.53, 90% CI 2-sided [98.60 to 104.54] — AUC0-inf Test/Reference Ratio

ADVERSE EVENTS:
Time Frame: Eighteen days for each arm (Safety Surveillance Period).
Description: Safety population included all subjects who received at least one dose of intervention.
Arm/Group | Temodal | Dralitem
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temodal (N=16) | Dralitem (N=16)
Itchy Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Hyporexia (Metabolism and nutrition disorders) | 1 | 0
Leg Edema (Vascular disorders) | 1 | 0
Weakness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Loss of taste (Nervous system disorders) | 1 | 0
Adynamia (Nervous system disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Expressive aphasia (Nervous system disorders) | 0 | 1
Fever syndrome (General disorders) | 0 | 1
Proctorrhagia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes